CLINICAL TRIAL: NCT06874322
Title: Voiceitt for People With Impairments in Speech
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Duquesne University (Other)
Responsible Party: Principal Investigator, Brad Dicianno, Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY24100164
Record Dates: First submitted 2025-02-21; First posted 2025-03-13 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Speech Impairment; Speech Disorder
Keywords: Speech Impairment; voice recognition tool; dictation tool; voice recognition app; dictation app; voiceitt app; speech disabilities; dysarthria; moderate dysarthria
MeSH Terms: conditions — Speech Disorders; Dysarthria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Voiceitt (Experimental): Participants will use Voiceitt App. Voiceitt is a voice recognition and dictation tool that adapts to users' unique, non-standard speech patterns. It integrates with mainstream devices and platforms to enable communication, accessibility, and independence for people with speech disabilities. https://www.voiceitt.com/
  Interventions: Other: Voiceitt

INTERVENTIONS:
Other: Voiceitt — Participants will use Voiceitt App

SUMMARY:
The primary objective of this pilot study is to evaluate the feasibility and preliminary effectiveness of the Voiceitt app in improving communication for individuals with speech impairments due to conditions such as cerebral palsy (CP), stroke, Amyotrophic Lateral Sclerosis (ALS), or Parkinson's disease.

DETAILED DESCRIPTION:
Conditions like CP, ALS, Stroke or Parkinson's disease, etc., cause communication impairment. There are few augmentative communication options that allow people with these impairments to communicate effectively.

Voiceitt is an app that is designed to assist people with speech impairments by using a voice recognition and dictation tool that adapts to users' unique, non-standard speech patterns. However, its effectiveness in clinical populations has not been established. This study is bridging the gap in evaluating the preliminary effectiveness and feasibility of Voiceitt app in improving communication among people with mild to moderate speech impairments.

ELIGIBILITY:
Inclusion Criteria:

* Age 13 or older
* moderately severe speech dysarthria due to conditions such as CP, stroke, ALS or Parkinson's Disease, etc.
* Ability to understand and follow instructions for using the Voiceitt app.

Exclusion Criteria:

* Severe cognitive impairments that prevent the understanding of the Voiceitt app and required training.
* Patients who have additional speech impairments other than dysarthria, such as significant aphasia or verbal apraxia.
* Severe physical impairments that prevent interaction with the app.
* Non-English speakers.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in Communication Abilities as measured by SIR | Baseline (Day 1), 5-6 months, and 7-8 months
  Change in Communication Abilities as measured by Speech Intelligibility Rating (SIR) that quantifies clarity of speech. The rating ranges from 1-5. low rating means speech is unintelligible, and highest rating means speech is intelligible to all listeners. Change in SIR is measured by administering SIR at 3 different time points, at baseline, and two times after intervention.
Change in Communication Abilities as measured by Communication Effectiveness Index (CETI) | Baseline (day 1), 5-6 months, and 7-8 months
  Change in Communication Abilities as measured by Communication Effectiveness Index (CETI) that measures perceived effectiveness of communication in daily activities. CETI is a 16 item questionnaire. Each item is scored from 1-100. The final score of CETI is the averaged score across the 16 items, and ranges from 1-100. A high score indicates good performance in functional communication and a low score, poor performance. Change in CETI is measured by administering CETI at 3 different time points, at baseline, and two times after intervention.

SECONDARY OUTCOMES:
User Satisfaction | 7-8 months
  User satisfaction is assessed through surveys and interviews focusing on ease of use, satisfaction with the app, and perceived changes. The survey uses Likert-type scale where users choose the answer option that represent their assessment of the app on several usability questions. An example of the question-and-answer choices is "How easy was it to set up the Voiceitt app? Very easy, Easy, Neutral, Difficult, Very difficult." Reported data will be a combination of frequency of participants choosing favorable and unfavorable answer choices, and a qualitative analysis based on participants' responses to the survey and interview.
Change in Communication-Related Frustration | 7-8 months
  Self-reported change in frustration levels during communication.
Change in Participants' Accounts on Social Interaction Quality | 7-8 months
  Through qualitative interviews, participants will be asked about how the app influenced their social interactions and participation in daily activities. This information will be reported qualitatively as themes using qualitative analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Brad E Dicianno, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Center for Assistive Technology, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No